CLINICAL TRIAL: NCT02895776
Title: Search for Risk Factors of Conversion From Local to General Sedation in Emergency Endovascular Therapy for Acute Stroke
Brief Title: Risk Factors of Conversion From Local to General Sedation in Endovascular Stroke Therapy
Acronym: AMAS
Status: Terminated | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: GTR_2015_23
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2017-09

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- General Sedation: Case patients: Endovascular Acute Stroke Therapy scheduled to be performed under local sedation and finally performed under General anesthesia
- local sedation: Control patients: Endovascular Acute Stroke Therapy scheduled to be performed, and actually performed under conscious Sedation

SUMMARY:
Thrombectomy is now the standard of care of revascularization in acute ischaemic stroke. Data tend to show that final neurologic outcome is superior if the thrombectomy procedure was performed under conscious sedation.

The Rothschild Foundation is a high output centre with more than 400 thrombectomy procedures every year.

We report a rate of 5% of these procedures requiring general anesthesia despite conscious sedation being the standard of care. This study aims to identify clinical factors associated with a risk of conversion of a conscious sedation to a general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thrombectomy for ischemic stroke
* age ≥ 18 years old

Exclusion Criteria:

* patient already under general anesthesia
* general sedation required
* haemorrhagic softening diagnosed before the beginning of procedure
* patient refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Endovascular Acute Stroke Therapy scheduled to be performed with local sedation and either performed under General Anesthesia (case), either actually performed under conscious sedation (control).
  Endovascular Acute Stroke Therapy scheduled to be performed with conscious sedation and performed under General Anesthesia 3 control patients will be included per case, and matched with the moment of procedure (term of the year).
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
factors associated with a conversion from conscious sedation to general anesthesia | during therapy (day 1)
  recording of the procedures during anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No